CLINICAL TRIAL: NCT04835688
Title: Transmyringeal Ventilation Tube Insertion for Unilateral Menière's Disease: a Prospective, Sham-controlled, Double-blinded, Randomized, Clinical Trial
Brief Title: Ventilation Tube Insertion for Unilateral Menière's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Casper Grønlund Larsen (Other)
Responsible Party: Sponsor-Investigator, Casper Grønlund Larsen, MD, PhD-student, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG1-2021
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-09

CONDITIONS: Meniere Disease
Keywords: Ventilation tube insertion; Grommet insertion; Vertigo
MeSH Terms: conditions — Meniere Disease; Vertigo | interventions — Middle Ear Ventilation

STUDY DESIGN:
Intervention Model Description: A pro-spective, double-blinded, sham-controlled, randomized, clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, care providers, data collectors, outcome assessors, research personnel, and data analysts will be blinded to treatment allocation. However, the ENT-specialist performing the insertion of the ventilation tube or placebo-treatment will inevitably be aware of treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilation tube insertion (Experimental): Ventilation tube insertion into the tympanic membrane.
  Interventions: Procedure: Transmyringeal ventilation tube insertion
- Sham-treatment (Sham Comparator): Sham-treatment. Manipulation of the tympanic membrane to simulate ventilation tube insertion without performing a ventilation tube insertion.
  Interventions: Procedure: Sham-treatment

INTERVENTIONS:
Procedure: Transmyringeal ventilation tube insertion — In both groups, the tympanic membrane will be anesthetized by local application of topical prilocaine (EMLA) or phenol or by infiltration anaesthesia of the outer ear canal. The choice of method is left to the discretion of the surgeon.
  For the experimental group, insertion of a ventilation tube will be performed. An incision is performed, usually in the lower, anterior quadrant of the tympanic membrane and the transmyringeal tube is inserted.
  Other Names: Ventilation tube insertion, grommet insertion
  Arms: Ventilation tube insertion
Procedure: Sham-treatment — For the control group, the ENT-specialist will touch the tympanic membrane with an alligator ear forceps to simulate getting a paracentesis. In the same procedure, without having made a paracentesis, a ventilation tube is placed on the tympanic membrane and removed again afterwards. The reason for the above-mentioned is to simulate getting a paracentesis and insertion of a ventilation tube.
  Arms: Sham-treatment

SUMMARY:
The purpose of this trial is to assess the effects of transmyringeal ventilation tubes compared with sham-treatment which do not ventilate the middle ear, on the number of vertigo attacks lasting more than 20 minutes in participants with Menière's disease.

DETAILED DESCRIPTION:
Menière's disease is an inner ear disorder with recurrent attacks of vertigo, fluctuating sensorineural hearing loss, tinnitus, and aural fullness. The underlying pathogenetic mechanisms are not known. The pathologic-anatomic correlate of the disease is endolymphatic hydrops, i.e. distension of the endolymphatic spaces as seen at post-mortem microscopic examination of the temporal bone. Prevalence-figures are in the range between 0.1% to 0.5% in the population. In Denmark, the estimated prevalence of Menière's disease is 3500. The disease commonly begins in the fourth or fifth decade of life, and the prevalence increases with age.

There are a great number of different treatment options for Menière's disease including diuretics, sodium-restriction, beta-histidine, and psycho-supportive means, most of which are not validated. The only validated treatment for the vertigo attacks is chemical labyrinthectomy by intra-tympanic injections of the ototoxic antibiotic gentamicin for which two double-blind, placebo-controlled trials found a significant effect. Treatment with gentamicin is ablative, i.e. the goal of the treatment is to destroy the vestibular sensors of the affected ear. This carries a risk of long-standing unsteadiness alongside with permanent hearing loss in the treated ear. Still, no treatments seem to protect from the hearing loss associated with Menière's disease.

The first to advocate the use of transmyringeal ventilation tubes for Menière's disease was Tumarkin in 1966. Tumarkin et al. suggested that negative middle-ear pressure, due to poor tubal function, would lead to a relative over-pressure in the inner ear and that this might be one of the mechanisms behind Menière's disease. In addition, Tumarkin et al. presented several cases where treatment with transmyringeal tubes resulted in relief from vertigo attacks. Hall and Brackmann performed tympanometry in patients with Menière's disease and showed that some, but not all, patients had negative middle-ear pressure and they questioned Tumarkin's suggestions.

ELIGIBILITY:
Inclusion Criteria:

Patients with definite or probable unilateral Menière's disease according to the diagnostic criteria formulated by the Classification Committee of the Bárány Society, The Japan Society for Equilibrium Research, the European Academy of Otology and Neurotology (EAONO), the Equilibrium Committee of the American Academy of Otolaryngology - Head and Neck Surgery (AAO-HNS), and the Korean Balance Society:

* Two or more spontaneous episodes of vertigo, each lasting 20 minutes to 12 hours
* Audiometrically documented low- to medium-frequency sensorineural hearing loss in the affected ear on at least one occasion before, during or after one of the episodes of vertigo
* Fluctuating aural symptoms (hearing, tinnitus or fullness) in the affected ear
* Not better accounted for by another vestibular diagnosis

Exclusion Criteria:

* Bilateral Menière's disease
* Additional neurotological disorders (e.g. vestibular migraine, vertebrobasilar transient ischemic attack or acoustic neuroma)
* Previous surgical therapy such as intratympanic gentamicin or endolymphatic sac surgery
* Expected problems to adhere to the study protocol (dementia, non-fluent in Danish, substance abuse, etc.)
* Previous treatment with transmyringeal ventilation tubes after childhood
* A serious illness that might interfere with treatment or follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of vertigo attacks lasting more than 20 minutes | 3 months
  Data will be collected as a patient-reported outcome by filling out a weekly self-evaluation of symptoms-questionnaire.
Number of vertigo attacks lasting more than 20 minutes | 24 months
  Data will be collected as a patient-reported outcome by filling out a weekly self-evaluation of symptoms-questionnaire.

SECONDARY OUTCOMES:
Pure-tone audiometry | 3 months
  4 tone average of 500, 1000, 2000, and 3000 Hz (dB) and 3 tone average of 125, 250, and 500 Hz (dB).
AAO-HNS Functional Level Scale | 3 months
  Questionnaire with written descriptions of how Menière's disease affects the life of the patient, from no impact at all to totally handicapped and unable to work.
Hearing, tinnitus, unsteadiness and aural fullness | 24 months
  Patient-reported outcome by filling out a self-evaluation of symptoms-questionnaire.
Number of subjects leaving | 24 months
  To check for unsatisfied treatment.
Number of subjects satisfied | 24 months
  To check for satisfied treatment
Speech audiometry | 3 months
  Discrimination in %.

CONTACTS AND LOCATIONS:
Overall Officials: Casper Grønlund Larsen, MD, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Køge, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data will be shared upon reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1/6-2024.
Access Criteria: Individual patient data will be shared upon reasonable request.

REFERENCES:
- [Derived] Larsen CG, Karlberg M, Guldfred F, Devantier L, Maagaard M, Homoe P, Djurhuus BD. Transmyringeal ventilation tube insertion for unilateral Meniere's disease: a protocol for a prospective, sham-controlled, double-blinded, randomized, clinical trial. Trials. 2022 Oct 17;23(1):877. doi: 10.1186/s13063-022-06777-w. PMID 36253829